CLINICAL TRIAL: NCT01762384
Title: Nationwide Multicenter Randomized Prospective Study to Compare Laparoscopic Sacral Colpopexy and Modified Total Pelvic Floor Reconstructive Surgery With Mesh for Apical Prolapse Stage III-IV
Brief Title: Laparoscopic Sacral Colpopexy Versus Modified Total Pelvic Floor Reconstructive Surgery for Apical Prolapse Stage III-IV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: pumch-gyn-05
Record Dates: First submitted 2012-12-30; First posted 2013-01-07 (Estimated); Last update posted 2013-01-07 (Estimated); Status verified 2012-12

CONDITIONS: Uterine Prolapse; Vault Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LSC (Active Comparator): procedure: laparoscopic sacral colpopexy.
  Interventions: Procedure: LSC; Device: "Gynemesh"
- Modified PFRS (Active Comparator): procedure: modified pelvic floor reconstructive surgery with mesh.
  Interventions: Procedure: modified PFRS; Device: "Gynemesh"

INTERVENTIONS:
Procedure: LSC — subjects of this group are submitted to surgical treatment of laparoscopic sacral colpopexy.
  Arms: LSC
Procedure: modified PFRS — subjects of this group are submitted to modified pelvic floor reconstructive surgery with mesh.
  Arms: Modified PFRS
Device: "Gynemesh" — Both surgeries will be conducted using mesh constructed from polypropylene mesh.

SUMMARY:
Pelvic Organ prolapse (a feeling of bulge in the vagina) may cause some distressing symptoms such as loss of control of the bowel or bladder, and may also cause problems with patient's sex life. The primary treatment is surgery. Sacral Colpopexy is the gold standard procedure. Now it could be done laparoscopically. Modified total pelvic floor reconstructive surgery with mesh is developed in China for Asian Women.

This study is designed to determine the effectiveness and safety of Modified total pelvic floor reconstructive surgery with mesh compared with laparoscopic Sacral Colpopexy for the treatment of uterine or vault prolapse Stage III-IV.

Patients enrolled into the study will be followed up for up to 3 years after surgery. Evaluation will take place during surgery and postoperative visit. Stage of prolapse before and after surgery, patient satisfaction through quality of life and sexual function questionnaires before and after surgery, and peri-operative complication rates will be evaluated.

DETAILED DESCRIPTION:
Pelvic organ prolapse is a common problem. The high rate of failure has led to an increasing use of synthetic grafts to augment vaginal repair procedures to obtain more durable results. In 2005, the investigators began to perform modified pelvic floor reconstruction surgery with mesh. The nation-wide multicenter prospective clinical trial data showed that it was safe, efficient and cost-effective. No severe intraoperative complications were recorded and the recurrence rate after 1 year follow-up was 8.1%. Quality of life improved significantly from the baseline, while the sexual function did not change.

Sacral colpopexy has long been regarded as the gold standard. Laparoscopic sacral colpopexy could offer durable result and low morbidity compared with open procedure.

In clinical practice, many women have symptomatic POP-Q Stage III-IV uterine or vault prolapse, which requires surgical correction. The aim of this multicenter, prospective and randomized study is to evaluate the effectiveness and safety of these two procedures in the treatment of symptomatic apical prolapse Stage III-IV in China.

ELIGIBILITY:
Inclusion Criteria:

* Candidates with symptomatic uterine or vault prolapse of Stage III-IV, suitable for surgical repair.
* Age from 55-65 years old.
* Agrees to participate in the study, including completion of all study-related procedures, evaluations and questionnaires.

Exclusion Criteria:

* Patients who could not tolerate laparoscopic surgery.
* Previous repair of pelvic organ prolapse involving insertion of mesh.
* Experimental drug or experimental medical device within 3 months prior to the planned procedure.
* Active genital, urinary or systemic infection at the time of the surgical procedure. Surgery may be delayed in such subjects until the infection is cleared.
* Coagulation disorder or on therapeutic anticoagulant therapy at the time of surgery.
* History of chemotherapy or pelvic radiation therapy. Systemic disease known to affect bladder or bowel function (e.g. Parkinson's disease, multiple sclerosis, spinal cord injury or trauma).
* Current evaluation or treatment for chronic pelvic pain (e.g. interstitial cystitis, endometriosis, coccydynia, vulvodynia).
* Nursing or pregnant or intends future pregnancy.
* Chronic cough not well-controlled.
* BMI ≥ 30.
* In the investigator's opinion, any medical condition or psychiatric illness that could potentially be life threatening or affect their ability to complete the study visits according to this protocol.

Ages: 55 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
anatomical improvement according to POP-Q score | 6 months
Anatomical improvement according to POP-Q Score | 1 year
Anatomical improvement according to POP-Q Score | 2 years
Anatomical improvement according to POP-Q Score | 3 years

SECONDARY OUTCOMES:
Hospital data:operative time | At discharge, an expected average of 5 days after operation.
Presence/absence of complications (composite score). | up to 6 weeks
  The occurrence (in the per-operative phase or within 6 weeks post-op) of at least one of the following: 1) bleeding complications; 2) infectious complications; 3) any wound caused by a surgeon movement: bladder, ureteral, or vascular injuries; 4)medical complications: deep vein thrombosis, pulmonary embolism and etc.Complications will be categorized using the Dindo surgical complication grading scale.
Change from baseline in PFIQ-7 scores. | 6 months, 1 year, 2 year, 3 year
Change from baseline in PFDI-21 scores. | 6 months, 1 year, 2 year, 3 year
In subjects sexually active at baseline, assessment of sexual function using PISQ-12 (mean scores and change from baseline) | 6 months, 1 year, 2 year, 3 year
Subject global impression assessed on a 5 point Likert scale | 6 months, 1 year, 2 year, 3 year
Presence/absence of complications (composite score) | up to 3 years
  Long-term negative outcomes of the surgical procedure will also be recorded until 3 years after surgery. For example, mesh erosion, de novo urinary incontinence, de novo dyspareunia and overall failure rate. Complications will be categorized using the Dindo surgical complication grading scale.
hospital data: estimated blood loss | At discharge, an expected average of 5 days after operation.
hospital data:length of stay | At discharge, an expected average of 5 days after operation.
hospital data: postoperative morbidity | At discharge, an expected average of 5 days after operation.
hospital data: time to recovery | At discharge, an expected average of 5 days after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Lan Zhu, Principal Investigator — Peking Union Medical College Hospital
Locations (4):
- China (4):
  - The First Affiliated Hospital of Guangzhou Medical College, Ghuangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang
  - Peking Union Medical College Hospital, Beijing